CLINICAL TRIAL: NCT00002198
Title: A Study to Investigate Whether There is a Pharmacokinetic Interaction Between 1592U89 and Ethanol Following Their Co-Administration to HIV-Infected Subjects.
Brief Title: A Study of 1592U89 and Ethanol When Given Together to HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 238F; CNAA 1010
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
Keywords: Drug Interactions; Antiviral Agents; Ethanol; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to see how the body processes 1592U89 and ethanol (pure grain alcohol) when they are given together.

DETAILED DESCRIPTION:
Patients are randomized to one of the following three regimens:

Regimen 1: 1592U89 alone. Regimen 2: pure grain alcohol diluted in orange juice. Regimen 3: 1592U89 plus pure grain alcohol diluted in orange juice. Treatment is administered weekly for 3 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Local treatment for Kaposi's sarcoma.
* Prophylactic treatment for opportunistic infections.

Patients must have:

* HIV-1 infection.
* CD4+ lymphocyte count >= 200 cells/microliter within 14 days prior to study drug administration.
* No active diagnosis of AIDS (other than visceral Kaposi's sarcoma) according to the 1993 Centers for Disease Control and Prevention (CDC) AIDS surveillance definition.

Prior Medication:

Allowed:

Local treatment for Kaposi's sarcoma.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

Malabsorption syndrome or other GI dysfunction which may interfere with drug absorption.

Concurrent Medication:

Excluded:

* Medications that cannot be withheld for 48 hours (24 hours for antiretrovirals) prior to study drug administration and until 12 hours after study drug administration on each dosing day.
* Immunomodulators, such as systemic corticosteroids, interleukins and interferons.
* Cytotoxic chemotherapeutic agents.
* Acute treatment for opportunistic infections.

Concurrent Treatment:

Excluded:

Radiation therapy.

Patients with the following prior conditions are excluded:

* Documented history of alcoholism.
* History of clinically relevant hepatitis or pancreatitis within 6 months prior to study drug administration.
* History of hypersensitivity, anaphylactic, or idiosyncratic reaction to nucleoside analogs.
* Participation in another research study within the past month.

Prior Medication:

Excluded:

* Cytotoxic chemotherapeutic agents within six weeks prior to study drug administration.
* Immunomodulating agents within six weeks prior to study drug administration.
* Treatment with the following within 2 weeks prior to study drug administration:
* acyclovir, carbamazepine, chloramphenicol, ganciclovir, phenytoin, rifampin, sodium valproate, or valacyclovir.

Prior Treatment:

Excluded:

Radiation therapy within 6 weeks prior to study drug administration.

1. Regular weekly alcohol intake of more than 21 units (a unit is equal to 1/2 pint beer or 1 glass of wine or 1 oz of liquor).

* Recent change in normal pattern of alcohol usage (e.g., prolonged use followed by > one month abstinence).
* Total abstinence from alcohol use.
* Positive breath alcohol test upon arrival at the study center prior to any dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, Inc, Wilmington, North Carolina, United States